CLINICAL TRIAL: NCT05358340
Title: Combined Spin- and Gradient-Echo Perfusion Weighted Imaging for Characterizing Vascular Architecture of Brain Lesions
Brief Title: Dual Perfusion Imaging for Characterizing Vascular Architecture of Brain Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-6282
Record Dates: First submitted 2022-04-26; First posted 2022-05-03 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Brain Tumor; Brain Metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — Perfusion Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (DSC MRI) (Experimental)
  Interventions: Diagnostic Test: Dynamic susceptibility contrast magnetic resonance imaging (DSC MRI)

INTERVENTIONS:
Diagnostic Test: Dynamic susceptibility contrast magnetic resonance imaging (DSC MRI) — A dye, known as a contrast agent, will be injected through a needle that is inserted into a vein in the arm or hand. Subsequent magnetic resonance imaging will follow.

SUMMARY:
The objectives of the study are (1) to evaluate the feasibility of using a combined spin- and gradient- echo (SAGE) sequence in dynamic susceptibility contrast magnetic resonance imaging (DSC MRI) and (2) to determine quantitative estimates of vessel density and size to differentiate between areas of radiation necrosis and tumor recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a brain metastasis or primary brain tumour and who will undergo MRI with contrast.

Exclusion Criteria:

* Subject or subject's legally authorized representative is unable or unwilling to consent to the study.
* Subject with documented contrast medium injection contraindication due to severe kidney disease or allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-24 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Measurement of perfusion parameter: cerebral blood volume (CBV) | Baseline to end of study (up to 2 years)
  Measurements of cerebral blood volume (CBV) will be calculated.
Measurement of perfusion parameter: vessel size index (VSI) | Baseline to end of study (up to 2 years)
  Measurements of vessel size index (VSI) will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Alcaide-Leon, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada